CLINICAL TRIAL: NCT05560841
Title: Prospective, " Evaluator Blinded " Clinical Investigation to Evaluate the Effectiveness and Safety of Nailner Brush 2-in-1 in the Treatment of Onychomycosis
Brief Title: Effectiveness and Safety of Nailner Brush 2in1 in Onychomycosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karo Pharma AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21E4142
Record Dates: First submitted 2022-09-15; First posted 2022-09-29 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Onychomycosis
MeSH Terms: conditions — Onychomycosis | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Topical application of Nailner brush 2in1 (medical device) for the treatment of toenail onychomycosis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nailner 2 in 1 (Experimental): Nailner Brush 2-in-1 (5ml)
  Liquid solution in glass bottle with a brush applicator Topical application twice a day during 4 weeks then once a day until 6 months
  Interventions: Device: topical treatment

INTERVENTIONS:
Device: topical treatment — Topical application of Nailner brush 2in1 for toenail onychomycosis

SUMMARY:
Evaluate the effectiveness of Nailner Brush 2-in-1 in the treatment of onychomycosis based on the blinded evaluation of the percentage of healthy nail surface after 6 months of treatment compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Patient having given freely her/his informed, written consent.
* Patient having a good general health.
* Age: between 18 and 70 years.
* Patient with superficial onychomycosis or light to moderate distolateral onychomycosis (without matrix involvement and involvement from 10 to 60%) on at least one great toenail.
* Patient with positive KOH staining.
* Patient cooperative and aware of the device modalities of use and the necessity and duration of the controls so that perfect adhesion to the protocol can be expected.
* Patient being psychologically able to understand information and to give their/his/her consent.
* Patient who agrees to refrain from receiving pedicure, artificial nails and/or cosmetic nail varnish or other medication on the nail being treated for the entire study duration.
* Female of childbearing potential should use a contraceptive regimen recognized as effective since at least 4 weeks before screening visit and during all the study.

Exclusion Criteria:

* Pregnant, breastfeeding woman or woman planning a pregnancy during the study;
* Patient enrolled in another clinical trial or which exclusion period is not over.
* Patient having used any systemic antifungal treatment in the last 6 months before screening and/or any topical antifungal treatment in the last months before screening visit.
* Patient with a condition or receiving a medication which, in the investigator's judgment, put the patient at undue risk;
* Patient suffering from a severe or progressive disease (at investigator's discretion) such as uncontrolled diabetes, peripheral circulatory disease, poor blood circulation HIV, psoriasis, lichen planus, immunosuppressive pathology, moderate and high risk obesity (BMI ≥30);
* Patient having a known allergy or hypersensitivity to one of the constituents of the investigational device.
* Patient with cutaneous pathology on studied zone (other than onychomycosis like angioma, dermatitis…).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the effectiveness of Nailner Brush 2-in-1 in the treatment of onychomycosis based on the blinded evaluation of the percentage of healthy nail surface after 6 months of treatment compared to baseline | Day 180
  Mean variation from baseline of the percentage of healthy surface after 6 months of treatment. Evaluation is done in blind by digital analysis of photographs of the infected toenail.

SECONDARY OUTCOMES:
To evaluate the effectiveness of Nailner Brush 2-in-1 in the treatment of onychomycosis based on the blinded evaluation of the percentage of healthy nail surface after 1 and 3 months of treatment compared to baseline | Day 30, Day 90
  Mean variation from baseline of the percentage of healthy surface after 1 and 3 months of treatment. Evaluation is done in blind by digital analysis of photographs of the infected toenail.
To evaluate the effectiveness of Nailner Brush 2-in-1 in the treatment of onychomycosis based on the microbiological cure (KOH staining) | Day 90, Day 180
  Percentage of patients with positive KOH staining at baseline and 3 and 6 months after treatment.
To evaluate the effectiveness of Nailner Brush 2-in-1 in the nail appearance | Day 30, Day 90, Day180
  Mean variation from baseline of the onychomycosis evaluation ( onycholysis, nail dystrophy, nail discoloration and nail thickening) as assessed by the investigator in live at baseline and 1, 3 and 6 months after treatment.
To evaluate the effectiveness of Nailner Brush 2-in-1 in the improvement of the quality of life (QoL) of the patients. | Day 7, Day 30, Day 90, Day 180
  Percentage of patient with an improvement of their quality of life (QoL) by analysis of NailQoL p
To evaluate the patient's opinion of Nailner Brush 2-in-1 effectiveness, tolerance, and acceptability. | Day 30, Day 90, Day 180
  Analysis of the answers to the patient questionnaire regarding effectiveness, tolerance, and acceptability of the investigational device 1, 3 and 6 months after treatment
To evaluate the safety of of Nailner Brush 2-in-1 | Day 180
  Product safety will be assessed by collection of Adverse Events (Aes) throughout the study. AEs will be summarized and tabulated by severity, causality, action taken and outcome, using descriptive statistics

CONTACTS AND LOCATIONS:
Overall Officials: Pr. Nejib DOSS, MD, Principal Investigator — Dermascan
Locations (2):
- Tunisia (2):
  - Private practice, Ben Arous
  - Private Practice, Tunis

IPD SHARING:
Plan to Share IPD: No